CLINICAL TRIAL: NCT00104702
Title: Radio-Surgical Treatment of Breast Cancer of Women Aged Over 70: Phase II Trial of Feasibility and Reproducibility of a Concentrated and Focalized Radiotherapy
Brief Title: Radiation Therapy in Treating Older Women Who Are Undergoing Surgery for Stage I or Stage II Breast Cancer
Acronym: GERICO03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000416123; FRE-FNCLCC-GERICO-03/0303; EU-20501
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemotherapy, Adjuvant; Radiotherapy

ARMS (1):
- Concentrated and Focalized Radiotherapy (Experimental)
  Interventions: Procedure: adjuvant therapy; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well radiation therapy works in treating older women who are undergoing surgery for stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine reproducibility of localized and concentrated adjuvant radiotherapy, in terms of isodose curve and dose heterogeneity, in older women with stage I or II breast cancer.

Secondary

* Determine the impact of this regimen on Katz's Activity of Daily Living score and Lawton's Instrumental Activity of Daily Living score in these patients.
* Determine relapse-free survival of patients treated with this regimen.
* Determine overall and specific survival of patients treated with this regimen.
* Determine the cosmetic result, as assessed by the patient, surgeon, and radiologist, of this regimen in these patients.
* Determine the direct and indirect costs of this regimen in these patients.

OUTLINE: This is a multicenter, open-label, nonrandomized study.

Patients undergo surgery. After surgery, patients undergo radiotherapy twice daily for 5 days.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of invasive breast cancer

  * Stage I or II disease

    * Tumor size ≤ 30 mm

      * Located in any breast quadrant
    * No nodal involvement
* No inflammatory breast cancer
* No positive margins after surgical resection (performed on study)
* No microcalcifications
* Hormone receptor status

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 70

Sex

* Female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-07; Primary Completion 2008-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Reproducibility | 1 month

SECONDARY OUTCOMES:
Impact of localized and concentrated radiotherapy on Katz's Activity of Daily Living score and Lawton's Instrumental Activity of Daily Living score | 3 weeks
Relapse-free survival | 1 year
Overall and specific survival | 1 year
Cosmetic result | 1 year
Direct and indirect costs | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: J. M. Hannoun-Levi, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (10):
- France (10):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Paul Strauss, Strasbourg
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif